CLINICAL TRIAL: NCT03535155
Title: Automated Spinal Landmark Identification to Improve Patient Safety and Efficacy During Neuraxial Anaesthesia Needle Insertion
Brief Title: Ultrasound Identification Automation Study
Status: Active, not recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: SHF-NHIC/MT006/2015
Record Dates: First submitted 2018-05-13; First posted 2018-05-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Spinal Anesthesia
Keywords: Ultrasound image, Neuraxial anesthesia, Landmark

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim of this study is to develop an automated spinal landmark identification system to improve patient safety and efficacy of neuraxial procedure needle insertion success.

This is a prospective cohort study to evaluate the accuracy of the automated spinal landmark identification technique using image processing system based on identification by experienced investigator using ultrasound in subjects requiring spinal anesthesia.

DETAILED DESCRIPTION:
Neuraxial procedures are commonly performed with wide range of therapeutic and diagnostic indications. Applications include neuraxial anesthesia for surgery, epidural labour analgesia, epidural steroid injections and lumbar punctures. The current blind palpation landmark technique is known to be highly inaccurate and may increase the risk of multiple insertion attempts, patient suffering and complication rates such as spinal cord injury. A key challenge for neuraxial procedures is the correct identification of needle insertion site.

The ultrasound imaging technique has found its way to neuraxial procedures as an imaging method to detect the inner anatomical structure of the lumbar spine and is superior to the traditional palpation method. However, a full interpretation of ultrasound images requires professional training and experience.

The overall aim of this proposal is to develop an automated spinal landmark identification system to improve patient safety and efficacy of neuraxial procedure needle insertion success. The primary aim is to develop an automated spinal landmark identification algorithm using image processing system to achieve 90% 1st spinal needle success rate within 12 months. The investigators will recruit 100 subjects in a prospective cohort study to investigate the spinal needle success rate as a clinically relevant outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21-75 years old who required spinal anesthesia for surgical procedure;
* Weight of 40-90kg and height of 140-180cm;
* BMI less than 30.

Exclusion Criteria:

* History of scoliosis;
* History of spinal instrumentation;
* Drug allergy to ultrasound transmission gel;
* Visible wound or injury in the lumbar spine.

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The women whose age between 21-75 years old who required spinal anaesthesia for surgical procedure.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
First attempt success rate of spinal anaesthesia | 12 hours
  First attempt success rate of spinal anaesthesia

SECONDARY OUTCOMES:
Number of spinal attempts | 12 hours
  The number of attempts to achieve successful spinal anaesthesia
Time taken to identify the ligamentum flavum in the transverse view | 12 hours
  Time taken to identify the ligamentum flavum in the transverse view
Distance from skin to ligamentum flavum | 12 hours
  Distance from skin to ligamentum flavum

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, MBBS, MMED, Principal Investigator — KK Women's and Children's Hospital

REFERENCES:
- [Derived] Oh TT, Ikhsan M, Tan KK, Rehena S, Han NR, Sia ATH, Sng BL. A novel approach to neuraxial anesthesia: application of an automated ultrasound spinal landmark identification. BMC Anesthesiol. 2019 Apr 16;19(1):57. doi: 10.1186/s12871-019-0726-6. PMID 30991949